CLINICAL TRIAL: NCT07016672
Title: Efficacy of Therapy With Intra-articular Injections of PRP Compared With Therapy With Intra-articular Injections of HA, in Patients With Grade III or IV GONArthrosis: a Prospective Randomized Open-label Study
Brief Title: Efficacy of Therapy With PRP Injections Versus HA in Patients With Advanced Grade of GONArthrosis
Acronym: PAGONA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Collaborators: Fondation Apicil (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-CHITS-001; 2024-A00370-47 (Other: IdRCB)
Record Dates: First submitted 2025-05-27; First posted 2025-06-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Knee Osteoarthritis
Keywords: Pain; Functional impact; Platelet Rich Plasma; hyaluronic acid; Intra-articular injection; Advanced grade
MeSH Terms: conditions — Osteoarthritis, Knee; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HA Injections (Active Comparator): Group 1: HA injections (3 injections at 7-day intervals)
  Interventions: Procedure: intra-articular injection of HA
- PRP Injections (Experimental): Group 2: PRP injections (3 injections at 15-day intervals)
  Interventions: Procedure: intra-articular injection of PRP

INTERVENTIONS:
Procedure: intra-articular injection of HA — 3 injections at 7-day intervals
  Arms: HA Injections
Procedure: intra-articular injection of PRP — 3 injections at 15-day intervals
  Arms: PRP Injections

SUMMARY:
Gonarthrosis is a chronic pathology affecting the knee joint and tissues. It is characterized by progressive degeneration of articular cartilage, bone and surrounding structures. Diagnosis is based on clinical, biological and radiological criteria.

When knee osteoarthritis becomes symptomatic, it leads to pain associated with stiffness and functional discomfort, impacting on patients' quality of life. Patients become sedentary and isolated, which has cardiovascular and psychological consequences, with a proven excess mortality rate.

To date, there are no curative treatments for gonarthrosis. Available treatments are generally aimed at relieving pain, improving joint function and slowing disease progression. Therapeutic approaches most often combine non-pharmacological treatments such as dietary measures, regular physical activity and therapeutic education, with pharmacological treatments: paracetamol, non-steroidal anti-inflammatory drugs, opioids, intra-articular injections of corticosteroids, hyaluronic acid (HA), Platelet Rich Plasma (PRP)... If these are ineffective, particularly in advanced stages (grades III-IV), then surgery for prosthesis is necessary. However, surgery is not an option for all patients, particularly those with co-morbidities, the elderly or those who refuse it.

The osteoarthritis section of the French rheumatology society has drawn up recommendations, with a view to positioning these treatments, standardizing practices and improving the management of gonarthrosis patients in France. These point out that further studies are needed to validate the efficacy of certain treatments, notably intra-articular PRP injections, which are nevertheless widely used in current practice and defended by a consensus of French experts published in 2021. Indeed, the results of several therapeutic trials and meta-analyses already published show that its efficacy is often superior to that of HA, particularly in terms of symptom improvement and over a longer duration. In order to make the case for their use to learned societies, literature data must be enriched, particularly with regard to advanced stages of gonarthrosis, i.e. stages III-IV, which are the most painful. The aim is to propose an effective treatment to relieve the symptoms of patients for whom surgery is not an option.

DETAILED DESCRIPTION:
In the PAGONA project, the investigators intend to use validated tools (WOMAC questionnaire, EVA scale, EQ-5D-5L quality of life questionnaire) to compare the effect of intra-articular injections of PRP with those of HA on the functional impact of the disease in patients with symptomatic knee osteoarthritis of moderate to severe stages (III-IV), by following these patients for 12 months after their last injection. The investigators plan to conduct a randomized, open-label study at the "Unité de Médecine et de Traumatologie du Sport" (UMTS) at Hôpital Sainte Musse in Toulon, where gonarthrosis treatment using intra-articular injections of PRP and HA is standard practice.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years ;
2. MRI confirmed grade III or IV unilateral gonarthrosis ;
3. Pain ≥ 3/10 on the visual analogue scale (VAS);
4. Patient with a BMI < 35
5. Patient capable of giving consent prior to participation in the study;
6. Affiliated or entitled under a social security scheme.

Exclusion Criteria:

1. Non-steroidal anti-inflammatory drugs or corticosteroids taken in the 7 days prior to inclusion;
2. Local injection of hyaluronic acid in the 2 months prior to inclusion;
3. Local injection of PRP within 1 year prior to inclusion;
4. Local injection of corticosteroids within 5 months prior to inclusion;
5. Current anticoagulant treatment that cannot be stopped for the duration of the study;
6. Patient diagnosed with any type of cancer in the last 3 years;
7. Pregnant women, women in labour or breast-feeding women;
8. Patients under judicial protection (guardianship, curatorship, etc.) or safeguard of justice;
9. Any other reason which, in the opinion of the investigator, could interfere with the evaluation of the study objectives.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Functional impact | 3 months after the last intra-articular injection
  The functional impact of the gonarthrosis will be assessed by the global WOMAC score, before injections and 3 months after the last injection, compared with the same score before treatment in each treatment group.
  The questionnaire consists of 24 questions divided into 3 categories: pain, physical function and stiffness.
  Each category offers a possible score range of 0 to 20 for pain, 0 to 68 for physical function, and 0 to 8 for stiffness. The sum of the scores for the three categories gives the total WOMAC score.
  The higher the score, the greater the functional impact of the gonarthrosis.

SECONDARY OUTCOMES:
Functional impact | up to 12 months
  The functional impact of the gonarthrosis will be assessed by the global WOMAC score, before injections and at 6 and 12 months after the last injection, compared with the same score before treatment in each treatment group. Evaluation of the overall WOMAC score beyond 3 months, and in each component of the WOMAC score (pain, stiffness and functional discomfort).
  The questionnaire consists of 24 questions divided into 3 categories: pain, physical function and stiffness.
  Each category offers a possible score range of 0 to 20 for pain, 0 to 68 for physical function, and 0 to 8 for stiffness. The sum of the scores for the three categories gives the total WOMAC score.
  The higher the score, the greater the functional impact of the gonarthrosis.
Pain evaluation | up to 12 months
  The patient's pain will be assessed before the 1st injection, at 3 months, 6 months and 12 months after the last injection using a Digital Visual Scale.
  The Visual Digital Pain Scale is a self-assessment pain intensity scale. It is used to quantify the pain felt by patients and to monitor its evolution. It is scored using 11 numbers, ranging from 0 ("No pain") to 10 ("Maximum imaginable pain"). Patients are asked to choose the number corresponding to the intensity of their pain.
  This scale gives a score from 0 to 10 (0 to 10 cm).
Failure rate | up to 12 months
  Therapeutic failure, defined as recourse to surgery (knee prosthesis) and/or recourse to additional injections of PRP or HA to relieve the patient and/or the occurrence of an intra-articular infection, assessed up to 12 months after the last injection.
Quality of life evaluation | up to 12 months
  EQ-5D-5L quality of life questionnaire scores assessed before the 1st injection, at 3 months, 6 months and 12 months after the last injection.
  EQ-5D-5L scores range from -0.59 to 1, where 1 is the best possible health status.
Adverse events | up to 12 months
  Number and description of adverse events related to HA or PRP injections assessed at 3 months, 6 months and 12 months after the last injection.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Jacques Raymond, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (1):
- Centre Hospitalier Intercommunal de Toulon- La Seyne sur Mer - Hôpital Sainte Musse, Toulon, Var, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vincent P. Acide hyaluronique intra articulaire dans la gonarthrose: une etude long-terme, ouverte, de Phase IV, avec analyse detaillee par stade de Kellgren-Lawrence. Curr Ther Res Clin Exp. 2020 May 27;92:100588. doi: 10.1016/j.curtheres.2020.100588. eCollection 2020. PMID 32714470
- [Background] Papalia R, Torre G, Zampogna B, Vorini F, Grasso A, Denaro V. Sport activity as risk factor for early knee osteoarthritis. J Biol Regul Homeost Agents. 2019 Mar-Apr;33(2 Suppl. 1):29-37. XIX Congresso Nazionale S.I.C.O.O.P. Societa' Italiana Chirurghi Ortopedici Dell'ospedalita' Privata Accreditata. PMID 31169000
- [Background] Sellam J, Courties A, Eymard F, Ferrero S, Latourte A, Ornetti P, Bannwarth B, Baumann L, Berenbaum F, Chevalier X, Ea HK, Fabre MC, Forestier R, Grange L, Lellouche H, Maillet J, Mainard D, Perrot S, Rannou F, Rat AC, Roux CH, Senbel E, Richette P; French Society of Rheumatology. Recommendations of the French Society of Rheumatology on pharmacological treatment of knee osteoarthritis. Joint Bone Spine. 2020 Dec;87(6):548-555. doi: 10.1016/j.jbspin.2020.09.004. Epub 2020 Sep 12. PMID 32931933
- [Background] Nuesch E, Dieppe P, Reichenbach S, Williams S, Iff S, Juni P. All cause and disease specific mortality in patients with knee or hip osteoarthritis: population based cohort study. BMJ. 2011 Mar 8;342:d1165. doi: 10.1136/bmj.d1165. PMID 21385807
- [Background] Altman R, Asch E, Bloch D, Bole G, Borenstein D, Brandt K, Christy W, Cooke TD, Greenwald R, Hochberg M, et al. Development of criteria for the classification and reporting of osteoarthritis. Classification of osteoarthritis of the knee. Diagnostic and Therapeutic Criteria Committee of the American Rheumatism Association. Arthritis Rheum. 1986 Aug;29(8):1039-49. doi: 10.1002/art.1780290816. PMID 3741515
- [Background] Bellamy N, Buchanan WW, Goldsmith CH, Campbell J, Stitt LW. Validation study of WOMAC: a health status instrument for measuring clinically important patient relevant outcomes to antirheumatic drug therapy in patients with osteoarthritis of the hip or knee. J Rheumatol. 1988 Dec;15(12):1833-40. PMID 3068365
- [Background] Zheng H, Chen C. Body mass index and risk of knee osteoarthritis: systematic review and meta-analysis of prospective studies. BMJ Open. 2015 Dec 11;5(12):e007568. doi: 10.1136/bmjopen-2014-007568. PMID 26656979
- [Background] Eymard F, Ornetti P, Maillet J, Noel E, Adam P, Legre-Boyer V, Boyer T, Allali F, Gremeaux V, Kaux JF, Louati K, Lamontagne M, Michel F, Richette P, Bard H; GRIP (Groupe de Recherche sur les Injections de PRP, PRP Injection Research Group). Intra-articular injections of platelet-rich plasma in symptomatic knee osteoarthritis: a consensus statement from French-speaking experts. Knee Surg Sports Traumatol Arthrosc. 2021 Oct;29(10):3195-3210. doi: 10.1007/s00167-020-06102-5. Epub 2020 Jun 24. PMID 32583023
- [Background] Alcerro JC, Lavernia CJ. Stem Cells and Platelet-rich Plasma for Knee Osteoarthritis: Prevalence and Cost in South Florida. J Am Acad Orthop Surg. 2019 Oct 15;27(20):779-783. doi: 10.5435/JAAOS-D-18-00343. PMID 30499895
- [Background] McElheny K, Toresdahl B, Ling D, Mages K, Asif I. Comparative Effectiveness of Alternative Dosing Regimens of Hyaluronic Acid Injections for Knee Osteoarthritis: A Systematic Review. Sports Health. 2019 Sep/Oct;11(5):461-466. doi: 10.1177/1941738119861545. Epub 2019 Jul 24. PMID 31340715
- [Background] Chu CR, Rodeo S, Bhutani N, Goodrich LR, Huard J, Irrgang J, LaPrade RF, Lattermann C, Lu Y, Mandelbaum B, Mao J, McIntyre L, Mishra A, Muschler GF, Piuzzi NS, Potter H, Spindler K, Tokish JM, Tuan R, Zaslav K, Maloney W. Optimizing Clinical Use of Biologics in Orthopaedic Surgery: Consensus Recommendations From the 2018 AAOS/NIH U-13 Conference. J Am Acad Orthop Surg. 2019 Jan 15;27(2):e50-e63. doi: 10.5435/JAAOS-D-18-00305. PMID 30300216
- [Background] Gormeli G, Gormeli CA, Ataoglu B, Colak C, Aslanturk O, Ertem K. Multiple PRP injections are more effective than single injections and hyaluronic acid in knees with early osteoarthritis: a randomized, double-blind, placebo-controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Mar;25(3):958-965. doi: 10.1007/s00167-015-3705-6. Epub 2015 Aug 2. PMID 26233594
- [Background] Lin KY, Yang CC, Hsu CJ, Yeh ML, Renn JH. Intra-articular Injection of Platelet-Rich Plasma Is Superior to Hyaluronic Acid or Saline Solution in the Treatment of Mild to Moderate Knee Osteoarthritis: A Randomized, Double-Blind, Triple-Parallel, Placebo-Controlled Clinical Trial. Arthroscopy. 2019 Jan;35(1):106-117. doi: 10.1016/j.arthro.2018.06.035. PMID 30611335
- [Background] Patel S, Dhillon MS, Aggarwal S, Marwaha N, Jain A. Treatment with platelet-rich plasma is more effective than placebo for knee osteoarthritis: a prospective, double-blind, randomized trial. Am J Sports Med. 2013 Feb;41(2):356-64. doi: 10.1177/0363546512471299. Epub 2013 Jan 8. PMID 23299850
- [Background] Smith PA. Intra-articular Autologous Conditioned Plasma Injections Provide Safe and Efficacious Treatment for Knee Osteoarthritis: An FDA-Sanctioned, Randomized, Double-blind, Placebo-controlled Clinical Trial. Am J Sports Med. 2016 Apr;44(4):884-91. doi: 10.1177/0363546515624678. Epub 2016 Feb 1. PMID 26831629
- [Background] Buendia-Lopez D, Medina-Quiros M, Fernandez-Villacanas Marin MA. Clinical and radiographic comparison of a single LP-PRP injection, a single hyaluronic acid injection and daily NSAID administration with a 52-week follow-up: a randomized controlled trial. J Orthop Traumatol. 2018 Aug 20;19(1):3. doi: 10.1186/s10195-018-0501-3. PMID 30128934
- [Background] Cerza F, Carni S, Carcangiu A, Di Vavo I, Schiavilla V, Pecora A, De Biasi G, Ciuffreda M. Comparison between hyaluronic acid and platelet-rich plasma, intra-articular infiltration in the treatment of gonarthrosis. Am J Sports Med. 2012 Dec;40(12):2822-7. doi: 10.1177/0363546512461902. Epub 2012 Oct 25. PMID 23104611
- [Background] Cole BJ, Karas V, Hussey K, Pilz K, Fortier LA. Hyaluronic Acid Versus Platelet-Rich Plasma: A Prospective, Double-Blind Randomized Controlled Trial Comparing Clinical Outcomes and Effects on Intra-articular Biology for the Treatment of Knee Osteoarthritis. Am J Sports Med. 2017 Feb;45(2):339-346. doi: 10.1177/0363546516665809. Epub 2016 Oct 21. PMID 28146403
- [Background] Di Martino A, Di Matteo B, Papio T, Tentoni F, Selleri F, Cenacchi A, Kon E, Filardo G. Platelet-Rich Plasma Versus Hyaluronic Acid Injections for the Treatment of Knee Osteoarthritis: Results at 5 Years of a Double-Blind, Randomized Controlled Trial. Am J Sports Med. 2019 Feb;47(2):347-354. doi: 10.1177/0363546518814532. Epub 2018 Dec 13. PMID 30545242
- [Background] Filardo G, Di Matteo B, Di Martino A, Merli ML, Cenacchi A, Fornasari P, Marcacci M, Kon E. Platelet-Rich Plasma Intra-articular Knee Injections Show No Superiority Versus Viscosupplementation: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1575-82. doi: 10.1177/0363546515582027. Epub 2015 May 7. PMID 25952818
- [Background] Huang Y, Liu X, Xu X, Liu J. Intra-articular injections of platelet-rich plasma, hyaluronic acid or corticosteroids for knee osteoarthritis : A prospective randomized controlled study. Orthopade. 2019 Mar;48(3):239-247. doi: 10.1007/s00132-018-03659-5. PMID 30623236
- [Background] Raeissadat SA, Rayegani SM, Ahangar AG, Abadi PH, Mojgani P, Ahangar OG. Efficacy of Intra-articular Injection of a Newly Developed Plasma Rich in Growth Factor (PRGF) Versus Hyaluronic Acid on Pain and Function of Patients with Knee Osteoarthritis: A Single-Blinded Randomized Clinical Trial. Clin Med Insights Arthritis Musculoskelet Disord. 2017 Oct 10;10:1179544117733452. doi: 10.1177/1179544117733452. eCollection 2017. PMID 29051707
- [Background] Su K, Bai Y, Wang J, Zhang H, Liu H, Ma S. Comparison of hyaluronic acid and PRP intra-articular injection with combined intra-articular and intraosseous PRP injections to treat patients with knee osteoarthritis. Clin Rheumatol. 2018 May;37(5):1341-1350. doi: 10.1007/s10067-018-3985-6. Epub 2018 Jan 31. PMID 29388085
- [Background] Dulic O, Rasovic P, Lalic I, Kecojevic V, Gavrilovic G, Abazovic D, Maric D, Miskulin M, Bumbasirevic M. Bone Marrow Aspirate Concentrate versus Platelet Rich Plasma or Hyaluronic Acid for the Treatment of Knee Osteoarthritis. Medicina (Kaunas). 2021 Nov 2;57(11):1193. doi: 10.3390/medicina57111193. PMID 34833411
- [Background] Joshi Jubert N, Rodriguez L, Reverte-Vinaixa MM, Navarro A. Platelet-Rich Plasma Injections for Advanced Knee Osteoarthritis: A Prospective, Randomized, Double-Blinded Clinical Trial. Orthop J Sports Med. 2017 Feb 13;5(2):2325967116689386. doi: 10.1177/2325967116689386. eCollection 2017 Feb. PMID 28255569
- [Background] Andrade LF, Ludwig K, Goni JMR, Oppe M, de Pouvourville G. A French Value Set for the EQ-5D-5L. Pharmacoeconomics. 2020 Apr;38(4):413-425. doi: 10.1007/s40273-019-00876-4. PMID 31912325
- See also: Related Info — https://www.ch-bourges.fr/wp-content/uploads/2022/04/Doc-PRP_site-Internet_v4.pdf
- See also: Related Info — https://www.has-sante.fr/upload/docs/application/pdf/2022-08/fiche_aps_arthroses_vf.pdf
- See also: Moustafa Naja. Stratégies de prise en charge de l'arthrose de genou : innovation et évaluation médico-économique. Médecine humaine et pathologie. Université de Strasbourg, 2022. Français. ⟨NNT : 2022STRAJ031⟩. ⟨tel-04008823⟩ — https://theses.hal.science/tel-04008823
- See also: Related Info — https://www.arthrolink.com/fr/dossiers-arthrose/tous-les-dossiers/arthrose-qualite-de-vie
- See also: Clark, Gregory P. DMSc, MPAS, PA-C. Treatment options for symptomatic knee osteoarthritis in adults. JAAPA 36(11):p 1-6, November 2023. — https://doi.org/10.1097/01.jaa.0000979536.73946.98